CLINICAL TRIAL: NCT04260477
Title: Novel Triple-dose Tuberculosis Retreatment Regimen: How to Overcome Resistance Without Creating More in Niger
Brief Title: Novel Triple-dose Tuberculosis Retreatment Regimen
Acronym: Tri-Do-Re
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Damien Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITM202001
Record Dates: First submitted 2020-02-03; First posted 2020-02-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Multidrug-resistant Tuberculosis; Pulmonary Tuberculosis; Tuberculosis; Resistance to Tuberculostatic Drugs
Keywords: rifampicin-susceptible-TB; Tuberculosis; first-line; TB relapse; TB treatment failure; high dose retreatment
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis, Pulmonary; Tuberculosis | interventions — Ethambutol; Isoniazid; Rifampin; Pyrazinamide

STUDY DESIGN:
Masking Description: Providers in the TB clinics and lab technicians in the Niger clinics and labs will not be blinded to the prescribed regimen. However, lab technicians working in the Institute of Tropical Medicine (ITM) lab will be blinded to the prescribed regimen. Also the statistician will be blinded to the prescribed regimen until the first interim analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6EH³R3Z (Experimental): (Rifampicin (R)/ Isoniazid (H) / Pyrazinamide (Z)/Ethambutol (E)) 6-month high-dose treatment; New high-dose isoniazid / high-dose rifampicin retreatment regimen (6EH³R3Z) - that includes triple-dose rifampicin (R3; 30 mg/kg), and triple-dose isoniazid (H3; 15 mg/kg), complemented with pyrazinamide (Z) and ethambutol (E).
  Interventions: Drug: 6EH³R³Z
- 6EHRZ (Active Comparator): Standard of care: 6-month 6RHZE regimen with dose combination tablets (one tablet: 150 mg R + 75 mg H + 400 mg Z + 275mg E)
  Interventions: Drug: 6EHRZ

INTERVENTIONS:
Drug: 6EH³R³Z — A triple dose is defined as the triple of the routine dose used for a specific WHO weight band. Hence, the mg/kg within a weigh-band varies, as is the case in routine practice.
  Dosing takings into consideration the fixed dose combination (FDC) tablets (one tablet: 150 mg R + 75 mg H + 400 mg Z + 275mg E). Dosage relies on tables with dosage by weight-bands used by WHO for the Cat. 1 regimen. The dosage used for the intensive phase of the Cat. 1 regimen applies for the whole treatment duration. A double dose of H and R is added to the recommended normal dose for adults (WHO,2003)
  Other Names: Ethambutol; isoniazid; rifampicin; pyrazinamide; triple dose isoniazid; triple dose rifampicin
  Arms: 6EH³R3Z
Drug: 6EHRZ — Recommended normal dose adults (WHO, 2003)
  * H: 5 (4-6) mg/kg/day
  * R: 10 (8-12) mg/kg/day
  * Z: 25 (20-30)mg/kg/day
  * E: 15 (15-18)mg/kg/day
  Other Names: Ethambutol; isoniazid; rifampicin; pyrazinamide
  Arms: 6EHRZ

SUMMARY:
To determine if a high-dose first-line regimen is non-inferior (non-inferiority margin 10%) in terms of safety to the same regimen at regular dosing, in previously treated patients with rifampicin-susceptible recurrent Tuberculosis (TB).

DETAILED DESCRIPTION:
Stage 1: This is a pragmatic open-label multi-stage randomized clinical trial. Potential participants will be screened and enrolled in Damien Foundation (DF) clinics participating in the trial.

First we will perform a two-arm study with 6EHRZ as control arm and 6EH³R³Z as intervention arm. If at interim analysis the intervention arm is not considered to be non-inferior to the control arm, the intervention stops and enrolment will continue in a an adapted intervention arm and the control arm (6EHRZ). Otherwise, enrolment continues to 6EHRZ and 6EH³R³Z.

Observational study (stage 2): The DSMB members agreed due to safety concerns to continuing the study as a cohort with only the control arm. The control regimen will remain the same (6EHRZ).

As per routine practice, during treatment patients are in daily contact with the direct observed therapy (DOT) supervisor and minimally monthly clinic visits are scheduled for monitoring of safety and treatment response.

Additionally, liver function tests will be performed at fixed intervals during treatment. Six month and one year after treatment completion or cure the patient will be checked for relapse with systematic sputum acid-fast bacilli (AFB)-microscopy and TB culture.

ELIGIBILITY:
Inclusion Criteria:

* All newly registered patients with smear-positive recurrent pulmonary TB
* Adults as well as children (no age limit)
* Able and willing to provide written informed consent
* Added for stage 2: lives within 5 km of a health facility with a medical doctor

Exclusion Criteria:

* All patients with TB initially resistant to rifampicin on Xpert MTB/RIF testing
* Patients transferred to a health facility not supported by the Damien Foundation
* Patients previously enrolled in the trial, and with another episode of rifampicin-susceptible TB during the study period
* Those with grade III elevation of liver function tests at baseline, or with clinically active liver disease at screening
* Pregnant or breastfeeding woman
* HIV co-infected patients requiring treatment with a protease inhibitor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
STAGE 1:number of patients with any grade 3-5 Adverse Event (AE) during treatment, assessed as probably or definitely related to TB treatment | 18 months
STAGE 2: Describe bacterial effectiveness | 18 months
  for stage 2 participants of the trial
STAGE 2: Describe acquired resistance | 18 months
  for stage 2 participants of the trial

SECONDARY OUTCOMES:
STAGE 1: number of previously treated patients with H-monoresistance and H-polyresistance, rifampicin (RMP) resistance missed by Xpert Mycobacterium tuberculosis (MTB)/rifampicin (RIF) | 18 months
  frequency of initial resistance patterns and mutations conferring resistance
STAGE 1: Programmatical effectiveness:number of participants with treatment success divided by number of participants with failure, death, or Lost to follow-up (LTFU) | 6 months, 18 months
  6 months treatment success: A patient with smear-positive Pulmonary Tuberculosis (PTB) at the beginning of treatment who completed treatment and sputum smear microscopy (SSM) negative in the last month of treatment and on at least one previous occasion or culture-negative at 6 months. A patient with smear-positive PTB at the beginning of treatment who completed treatment without clinical evidence of failure but with no record of sputum smear or culture results in the last month of treatment (either because tests were not done or because results are unavailable) 18 months treatment success: Those who were cured or completed treatment and were evaluated at 12 months post-treatment to be a) SSM negative , or b) SSM positive but culture (CU) negative, or c) without sputum and no clinical signs of TB.
STAGE 1: Clinical effectiveness: number of participants with treatment success, divided by number of participants with failure or death | 6 months, 18 months
  6 months treatment success: A patient with smear-positive PTB at the beginning of treatment who completed treatment and SSM negative in the last month of treatment and on at least one previous occasion or culture-negative at 6 months. A patient with smear-positive PTB at the beginning of treatment who completed treatment without clinical evidence of failure but with no record of sputum smear or culture results in the last month of treatment (either because tests were not done or because results are unavailable) 18 months treatment success: Those who were cured or completed treatment and were evaluated at 12 months post-treatment to be a) SSM negative , or b) SSM positive but CU negative, or c) without sputum and no clinical signs of TB.
STAGE 1:Bacteriological effectiveness : number of participants with treatment success, divided by number of participants with failure | 6 months, 18 months
  6 months treatment success: A patient with smear-positive PTB at the beginning of treatment who completed treatment and SSM negative in the last month of treatment and on at least one previous occasion or culture-negative at 6 months. A patient with smear-positive PTB at the beginning of treatment who completed treatment without clinical evidence of failure but with no record of sputum smear or culture results in the last month of treatment (either because tests were not done or because results are unavailable) 18 months treatment success: Those who were cured or completed treatment and were evaluated at 12 months post-treatment to be a) SSM negative , or b) SSM positive but CU negative, or c) without sputum and no clinical signs of TB.
STAGE 2:Bacteriological effectiveness : number of participants with treatment success, divided by number of participants with failure | 6 months, 18 months
  6 months treatment success: A patient with smear-positive PTB at the beginning of treatment who completed treatment and SSM negative in the last month of treatment and on at least one previous occasion or culture-negative at 6 months. A patient with smear-positive PTB at the beginning of treatment who completed treatment without clinical evidence of failure but with no record of sputum smear or culture results in the last month of treatment (either because tests were not done or because results are unavailable) 18 months treatment success: Those who were cured or completed treatment and were evaluated at 12 months post-treatment to be a) SSM negative , or b) SSM positive but CU negative, or c) without sputum and no clinical signs of TB.
STAGE 2: number of participants with acquired resistance, to Isoniazid (INH) and/or RMP | 6 months, 18 months
  In patients with recurrence, the recurrent strain will be compared with the diagnostic strain to identify possible differences in the resistance pattern. If the strain is the same, and resistance is not present in the diagnostic sample but is identified in the recurrence sample, then this resistance is considered as acquired. Resistance is defined as a) on genotypic Drug susceptibility testing (DST) (Deeplex or other): presence of a mutation in the resistance determining region for the drug with exception of generally recognized polymorphisms and silent mutations not leading to an error in the gene product. Heteroresistance at the proportion detectable by these methods will be considered at par with full-blown resistance, or b) growth at the critical concentration for the drug tested in phenotypic DST.
number of participants with stable (without reversion) SSM conversion | 2 months
  conversion to 0 AFB per field, without subsequent treatment failure
STAGE 1: number of participants with drug-induced hepatotoxicity | 18 months
  hepatotoxicity due to anti-TB drug treatment was defined as the following criteria:
  1. Grade 3-5 elevation of Liver function test (LFT), or grade 2 elevation of liver function tests with jaundice; AND
  2. absence of serological evidence of infection with hepatitis B or C, AND
  3. normalization or at least a 50% improvement in abnormal liver chemistry results after withdrawal of anti-TB drugs
STAGE 1:number of participants with any TB treatment change due to drug-induced hepatoxicity | 18 months
STAGE 1:number of participants with any TB treatment change due to AE | 18 months
STAGE 1:number of participants with any grade 3-5 AE | 18 months
STAGE 1:number of participants with any Serious Adverse Event (SAE) | 18 months
STAGE 2: number of participants with drug-induced hepatotoxicity | 18 months
  hepatotoxicity due to anti-TB drug treatment was defined as the following criteria:
  1. Grade 3-5 elevation of Liver function test (LFT), or grade 2 elevation of liver function tests with jaundice; AND
  2. absence of serological evidence of infection with hepatitis B or C, AND
  3. normalization or at least a 50% improvement in abnormal liver chemistry results after withdrawal of anti-TB drugs
STAGE 2:number of participants with any TB treatment change due to drug-induced hepatoxicity | 18 months
STAGE 2:number of participants with any TB treatment change due to AE | 18 months
STAGE 2:number of participants with any grade 3-5 AE | 18 months
STAGE 2:number of participants with any Serious Adverse Event (SAE) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sani Kadri, Principal Investigator — Ministry of Health, Niger
Locations (1):
- Damien Foundation, Niamey, Niger

IPD SHARING:
Plan to Share IPD: No